CLINICAL TRIAL: NCT02592655
Title: Randomized Sequence, Assessor-Blind, Cross-Over Study of a Windlass Tourniquet, a Pneumatic Tourniquet and an Elastic Adhesive Bandage for Use as a Tourniquet
Brief Title: A Transparent Elasticized Adhesive Occlusive Compression Bandage for Use as an Arterial Tourniquet
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Marcus Migura (Individual)
Collaborators: Mercy Health (Other)
Responsible Party: Sponsor-Investigator, Marcus Migura, Sponsor-Investigator, Migura, Marcus
Organization: Migura, Marcus (Individual)
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: HCT001
Record Dates: First submitted 2015-10-27; First posted 2015-10-30 (Estimated); Results first posted 2017-08-24 (Actual); Last update posted 2017-08-24 (Actual); Status verified 2016-01

CONDITIONS: Hemorrhage; Vascular Injury
Keywords: tourniquet; arterial; pre-hospital; SOFTT-W; Battle Wrap; windlass; exsanguination; hemorrhage; amputation
MeSH Terms: conditions — Hemorrhage; Vascular System Injuries; Exsanguination

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- Pneumatic Tourniquet (Active Comparator): All participants randomly allocated to receive all interventions. Pneumatic Tourniquet: The Automatic Tourniquet System (ATS) 1500 by Zimmer (formerly Aspen Labs) is a pneumatic tourniquet that is typically used in surgical settings, and is representative of best outcome under the ideal circumstances of a controlled environment. The 10 cm (4 inch) wide cylindrical cuff was used for all participants.
  Interventions: Device: Pneumatic Tourniquet
- Windlass Tourniquet (Active Comparator): Windlass Tourniquet with a 3.8 cm (1.5 inch) wide strap is representative of the typical use device in civilian prehospital and military combat environments. In accordance with current prehospital guidelines: If distal perfusion is observed after One Windlass Tourniquet is applied then a second windlass tourniquet will be applied immediately proximal to the first windlass tourniquet so that the participant has Two Windlass Tourniquets applied.
  Interventions: Device: One Windlass Tourniquet; Device: Two Windlass Tourniquets
- Tourniquet Tape 10 cm (Experimental): Tourniquet Tape 10 cm wide is a highly elastic transparent occlusive tape that is expected to create sufficient circumferential pressure to occlude arterial blood flow when tightly wrapped around a limb. The tape should be applied in mostly overlapping layers. The final wrap should be applied without tension to prevent the elastic tension from causing the tape to unwind itself.
  Interventions: Device: Tourniquet Tape 5 cm
- Tourniquet Tape 5 cm (Experimental): Tourniquet Tape 5 cm wide is a highly elastic transparent occlusive tape that is expected to create sufficient circumferential pressure to occlude arterial blood flow when tightly wrapped around a limb. The tape should be applied in mostly overlapping layers. The final wrap should be applied without tension to prevent the elastic tension from causing the tape to unwind itself.
  Interventions: Device: Tourniquet Tape 10 cm

INTERVENTIONS:
Device: Pneumatic Tourniquet — Automated pneumatic tourniquet, applied to middle upper thigh.
  Other Names: Zimmer Automatic Tourniquet System (ATS) 1500
  Arms: Pneumatic Tourniquet
Device: One Windlass Tourniquet — One Windlass Tourniquet 3.8 cm (1.5 inch) wide. A Special Operations Forces Tactical Tourniquet Wide (SOFTT-W) will be used for the windlass tourniquet. One windlass tourniquet will be applied to the middle upper thigh.
  Other Names: Special Operations Forces Tactical Tourniquet Wide (SOFTT-W)
  Arms: Windlass Tourniquet
Device: Two Windlass Tourniquets — Two Windlass Tourniquets will be applied by applying a second 3.8 cm (1.5 inch) wide windlass tourniquet immediately proximal to the first windlass tourniquet.
  Arms: Windlass Tourniquet
Device: Tourniquet Tape 5 cm — Tourniquet Tape is 5 cm (2 inch) in width. Tourniquet Tape is a highly elastic transparent occlusive material that can create circumferential pressure when stretched and wrapped around a limb. The tape should be stretched and overlapped by at least half the width as it is applied. The final wrap should be applied without tension.
  Arms: Tourniquet Tape 10 cm
Device: Tourniquet Tape 10 cm — Tourniquet Tape is 10 cm (4 inch) in width. Tourniquet Tape is a highly elastic transparent occlusive material that can create circumferential pressure when stretched and wrapped around a limb. The tape should be stretched and overlapped by at least half the width as it is applied. The final wrap should be applied without tension.
  Arms: Tourniquet Tape 5 cm

SUMMARY:
This cross-over study of twenty five (anticipated) healthy human subjects will utilize two active control devices, and two different widths of the investigational device. One active control is representative of the usual care tourniquet applied in hospital settings. The second active control is a windlass tourniquet representative of the pre-hospital and military usual care tourniquet device. Two inch and four inch widths of the investigational device will be evaluated. The purpose of this study is to characterize and compare investigational and control tourniquet safety and efficacy. All tourniquets will be applied to the upper thigh. Efficacy data is provided by the presence or absence of popliteal flow when assessed with ultrasound. Mapping of interface pressures between the skin and the tourniquet will provide safety data. A minimum washout of five minutes will be allowed between tourniquet applications. All interventions will be applied in one visit. No follow up visit is anticipated.

DETAILED DESCRIPTION:
This is a small study of 19 participants conducted over only two days. All data for this study is collected by the study.

Tourniquet application:

All tourniquet applications conducted with the participant seated on the edge of an exam table with one leg hanging off the side, and the leg for tourniquet application extended outward, with the mid calf resting on a support. This position permits access to the popliteal artery for ultrasonography while the investigator has access to apply the tourniquet. The lower edge of each tourniquet is aligned just above the middle of the thigh. All tourniquets are applied over the pressure mapping sensor. The sensor is slightly thicker than denim jeans. Extra care must be taken to ensure that the material of the sensor does not interfere with removing the slack from the windlass tourniquets before turning the windlass to apply final pressure.

When a second windlass tourniquet is to be applied it is applied just above or proximal to the first windlass tourniquet. The windlass of each tourniquet are located as far from each other as possible. Meaning that if the windlass of the first tourniquet is the twelve o'clock position then the windlass of the second tourniquet is positioned at the six o'clock position. The strap of each tourniquet cannot slip over the windlass of the other. This 6 and 12 positioning prevents the strap of the second windlass tourniquet from slipping over the first as it is tightened.

When the tape tourniquet is applied, it is elongated, stretched as it is layered over the preceding layer with at least one half over lap. The tape tourniquet used in this study is similar to, but not the same as the product called manufactured by Entrotech, called "Battle Wrap." Results similar to this study should not be expected with the "Battle Wrap" product.

ELIGIBILITY:
Inclusion Criteria:

1. Upper thigh circumference greater than 61 cm or 24 inches.
2. Upper thigh circumference greater than the 50th percentile based on available anthropometric data.

Exclusion Criteria:

1. Currently taking medications for the treatment of hypertension.
2. Cardiac, renal, pulmonary, hepatic or hemologic disease or disorder.
3. Patients with signs or symptoms of vascular insufficiency. Specifically, patients with any history of non-healing wound, ulcer, blood clots or peripheral vascular disease will be excluded.
4. Any coagulation disorder, prior thrombotic or embolic events such as a deep vein thrombosis.
5. Sickle cell.
6. Diabetes mellitus
7. Rheumatic arthritis or other auto immune disease.
8. Major surgery, significant traumatic injury, within 60 days trial.
9. Skin grafts on lower extremities.
10. Known or observed neurological symptoms, to include peripheral neurological symptoms or deficits.
11. Pregnant women, and women who suspect themselves to be pregnant are not eligible for this study.
12. Any known malignancy.
13. Claudication

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 19 (Actual)
Dates: Start 2015-12; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Marcus W Migura, Principal Investigator — Unafiliated
Locations (1):
- Vascular Medicine & Surgical Associates, Youngstown, Ohio, United States

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data will be de-identified and consolidated into one Excel file and made available online. Still ultrasound images used for primary outcome assessment will be consolidated into one pdf and made available online. Individual participant data that is not supported by clinicaltrials.gov will be posted with Zenodo or by other means. The intent to release de-identified data was disclosed to each volunteer during the informed consent process.
Supporting Information: ICF, CSR
Time Frame: Upon publication of summary results. Web links are provided in the references section.
Access Criteria: De-identified IPD from this study will be public domain. Identifying information and records will be held confidential.

REFERENCES:
- [Background] Kragh JF Jr, O'Neill ML, Walters TJ, Dubick MA, Baer DG, Wade CE, Holcomb JB, Blackbourne LH. The military emergency tourniquet program's lessons learned with devices and designs. Mil Med. 2011 Oct;176(10):1144-52. doi: 10.7205/milmed-d-11-00114. PMID 22128650
- [Background] Wenke JC, Walters TJ, Greydanus DJ, Pusateri AE, Convertino VA. Physiological evaluation of the U.S. Army one-handed tourniquet. Mil Med. 2005 Sep;170(9):776-81. doi: 10.7205/milmed.170.9.776. PMID 16261983
- [Background] Taylor DM, Vater GM, Parker PJ. An evaluation of two tourniquet systems for the control of prehospital lower limb hemorrhage. J Trauma. 2011 Sep;71(3):591-5. doi: 10.1097/TA.0b013e31820e0e41. PMID 21768905
- [Background] Swan KG Jr, Wright DS, Barbagiovanni SS, Swan BC, Swan KG. Tourniquets revisited. J Trauma. 2009 Mar;66(3):672-5. doi: 10.1097/TA.0b013e3181986959. PMID 19276736
- [Background] King RB, Filips D, Blitz S, Logsetty S. Evaluation of possible tourniquet systems for use in the Canadian Forces. J Trauma. 2006 May;60(5):1061-71. doi: 10.1097/01.ta.0000215429.94483.a7. PMID 16688072
- [Background] Walters TJ, Mabry RL. Issues related to the use of tourniquets on the battlefield. Mil Med. 2005 Sep;170(9):770-5. doi: 10.7205/milmed.170.9.770. PMID 16261982
- [Background] Walters TJ, Wenke JC, Kauvar DS, McManus JG, Holcomb JB, Baer DG. Effectiveness of self-applied tourniquets in human volunteers. Prehosp Emerg Care. 2005 Oct-Dec;9(4):416-22. doi: 10.1080/10903120500255123. PMID 16263675
- [Background] Ruterbusch VL, Swiergosz MJ, Montgomery LD, Hopper KW, Gerth WA. (U) ONR/MARCORSYSCOM Evaluation of Self-Applied Tourniquets for Combat Applications. Panama City, FL, US : Navy Experimental Diving Unit, November 10, 2005. NEDU Technical Report No.05-15.
- [Background] Hill JP, Montgomery LD, Hopper KW, Roy LA. (U) ONR/MARCORSYSCOM Evaluation of Self-Applied Tourniquets for Combat Applications, Second Phase. Panama City, FL, US : Navy Experimental Diving Unit, April 3, 2007. NEDU Technical Report No.07-07.
- [Background] Thomas J. Walters PhD; Joseph C. Wenke PhD; SFC Dominique; Greydanus, USA; David S. Kauvar MD, CPT, MC; David G. Baer PhD. (U) U. S. Army Institute of Surgical Research Laboratory Evaluation of Battlefield Tourniquets in Human Volunteers, Ft. Sam Houston, TX: U. S. Army Institute of Surgical Research, September 30, 2005. USAISR Technical Report No.2005-05
- Available data/document: Primary Outcome Ultrasound Images — https://doi.org/10.5281/zenodo.236263 — NCT02592655 Primary Outcome Tourniquet Study
- Available data/document: Individual Participant Data Set — https://doi.org/10.5281/zenodo.237773 — NCT02592655 Individual level data set
- Available data/document: Informed Consent Form — https://doi.org/10.5281/zenodo.245150 — Informed consent form containing description of study and procedures.

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Healthy volunteers with a minimum upper thigh circumference of 61 cm were recruited from the general population during the first two weeks of December 2015.
Pre-assignment Details: Each participant receives a different intervention each period. 19 Participants randomly allocated to unique sequences of four interventions. No participants were lost once enrolled. 5 minute minimum washout period between interventions.
Groups:
- All Participants: Each subject has been randomly allocated to a sequence of interventions. Pneumatic tourniquet with a 10 cm (4 inch) wide cylindrical cuff typically used in surgical settings, and is representative of best outcome.
  Windlass Tourniquet: The Special Operations Forces Tactical Tourniquet Wide (SOFTT-W) is 3.8 cm (1.5 inch) in width. The SOFTT-W is representative of the typical emergency tourniquet. In accordance with current prehospital guidelines: If a single windlass tourniquet not effective then a second windlass tourniquet will be applied immediately proximal to the first.
  Tourniquet Tape 10 cm wide and Tourniquet Tape 5 cm wide are elastic adhesive tape tourniquets.
  5 cm tape was discontinued after the 4th participant. Once stretched the tape was too narrow for sufficient overlap. Because the overlap was not sufficient the edges began to roll. This would create an unacceptably narrow band if left in place longer than the prescribed time.
Period: First Tourniquet, Left Thigh.
Arm/Group | All Participants
Started | 19
ATS (Pneumatic) | 5
Windlass Tourniquet | 7
Tourniquet Tape 10 cm Width | 5
Tourniquet Tape 5 cm Width | 2
Completed | 19
Not Completed | 0
Period: Second Tourniquet Right Thigh.
Arm/Group | All Participants
Started (Participants switch to different interventions each period.) | 19
ATS (Pneumatic) | 5
Windlass Tourniquet | 8
Tourniquet Tape 10 cm Width | 5
Tourniquet Tape 5 cm Width | 1
Completed | 19
Not Completed | 0
Period: Third Tourniquet, Left Thigh.
Arm/Group | All Participants
Started (Participants switch to different interventions each period.) | 19
ATS (Pneumatic) | 8
Windlass Tourniquet | 4
Tourniquet Tape 10 cm Width | 6
Tourniquet Tape 5 cm Width | 1
Completed | 19
Not Completed | 0
Period: Fourth Tourniquet Right Thigh.
Arm/Group | All Participants
Started (Investigator decided to discontinue the 5 cm Tourniquet Tape after the 4th participant.) | 4 (Only the first 4 participants received all four interventions.)
ATS (Pneumatic) | 1
Windlass Tourniquet | 0
Tourniquet Tape 10 cm Width | 3
Tourniquet Tape 5 cm Width | 0
Completed | 4
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: "One Windlass" indicates the participants received only one windlass tourniquet because it appeared to be effective. "Two Windlass" describes the participants that received two windlass tourniquets because one did not appear to be effective. The total describes all participants. All participants received both the pneumatic and tape tourniquet.
Groups:
- One Windlass Tourniquet: Baseline characteristics for participants that received only one windlass tourniquet.
- Two Windlass Tourniquets: Baseline characteristics for participants who had a second windlass tourniquet applied immediately proximal to the first. Meaning that a single windlass tourniquet did not appear effective.
- Total: Total of all reporting groups
Arm/Group | One Windlass Tourniquet | Two Windlass Tourniquets | Total
Number analyzed (Participants) | 8 | 11 | 19
Age, Continuous [Mean (Standard Deviation); unit: years] | 30.5 (9.5) | 36.1 (8.8) | 33.7 (9.25)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 4 | 4
  Male | 8 | 7 | 15
Body Mass Index (BMI) [Mean (Standard Deviation); unit: Kg/m^2] — Body Mass Index is the individual participants body weight in kilograms divided by the individual participants height in meters squared.
  Kg/m^2 | 27.4 (1.7) | 36.1 (4.3) | 32.4 (5.6)
BMI Weight Status Category (CDC) [Count of Participants; unit: Participants]
  BMI 18.5 - 24.9 Normal | 1 | 0 | 1
  BMI 25.0 - 29.9 Overweight | 7 | 1 | 8
  BMI 30.0 and Above Obese | 0 | 10 | 10
Weight [Mean (Standard Deviation); unit: kg] | 87.5 (11.0) | 111.3 (21.5) | 101.25 (21.22)
Height [Mean (Standard Deviation); unit: cm] | 178.6 (9.7) | 175.0 (10.1) | 176.5 (9.8)
Thigh Circumference [Mean (Standard Deviation); unit: cm] — All thigh circumference measures taken from the participants right thigh while standing.
  Upper thigh circumference: Measured just below the gluteal furrow.
  10 cm Above Mid Thigh: Circumference measured 10 cm above the mid point between the gluteal furrow and supra-patellar border.
  Middle thigh circumference: Circumference measured at the mid point between the gluteal furrow and the supra-patellar border.
  Lower Thigh: Circumference measured just above the supra-patellar border.
  cm
    Upper Thigh | 63.5 (3.7) | 71.2 (5.9) | 68.0 (6.3)
    10 cm above Mid Thigh | 61.0 (4.0) | 68.7 (5.7) | 65.4 (6.3)
    Middle Thigh | 55 (4.2) | 60.3 (5.3) | 58.1 (5.5)
    Lower Thigh | 42.3 (4.4) | 45.8 (3.1) | 44.3 (4.0)
Percentile of Mean Thigh Circumference [Number; unit: Percentile] — The mean thigh circumference for the specified set of participants has been compared to the 2010 ANTHROPOMETRIC SURVEY OF U.S. MARINE CORPS PERSONNEL: METHODS AND SUMMARY STATISTICS to determine the nth percentile rank reported. (see references)
  Percentile
    Upper thigh circumference percentile | 65 | 95 | 90
    Lower thigh circumference percentile | 75 | 95 | 90
Systolic Blood Pressure (SBP) [Mean (Standard Deviation); unit: mmHg] | 130 (8.8) | 136 (10.4) | 133 (10.0)
Limb Occlusion Pressure [Mean (Standard Deviation); unit: mmHg] — A 10 cm (4 inch) wide pneumatic tourniquet cuff was used with the Automatic Tourniquet System (ATS) 1500 by Aspen Labs to obtain Limb Occlusion Pressures (LOP) on the upper half of each participants thigh. Pulsatile flow was not observable for one sustained minute with duplex ultrasound at the popliteal artery.
  mmHg | 280 (30) | 319 (44) | 302 (43)
Ankle Brachial Index (ABI) [Mean (Standard Deviation); unit: Ratio] — For each participant the Ankle Brachial Index (ABI) was measured bilaterally, and the highest of the two were used to determine the mean and standard deviation for the specified group reported. An ABI less than 1.0 would be indicative of peripheral artery disease. An ABI greater than 1.4 would be indicative of an incompressible artery.
  Ratio | 1.15 (0.08) | 1.16 (0.11) | 1.16 (0.09)

OUTCOME MEASURES:

1. Primary Outcome: Radiologist Limb Occlusion Assessment
Description: Duplex and color flow ultrasound are used to assess distal blood flow at the popliteal artery for 1 sustained minute following the application of a each tourniquet intervention to the middle upper thigh. If no flow is observed for 1 sustained minute then it is considered successful occlusion. A still image is then saved for later evaluation by the blinded outcome assessor.
  The 5 cm tape was discontinued after the 4th participant because the tape was considered to unacceptably narrow after stretching and this was considered a mechanical failure even if occlusion was observed. Therefore the 5 cm tape data was not evaluated by the radiologist.
Time Frame: For 1 sustained minute after application of each tourniquet intervention.
Population: One ultrasound image from one of the participants of the pneumatic tourniquet (ATS) group failed to capture anatomy and was therefore not included in the analysis.
  One ultrasound image from one of the participants of the windlass tourniquet (SOFTT-W) group failed to capture anatomy and was therefore not included in the analysis.
Measure: Count of Participants; unit: Participants
Groups:
- Tourniquet Tape 10 cm: Tourniquet Tape 10 cm (4 inch) width. Duplex and color flow ultrasound are used to assess distal blood flow at the popliteal artery for 1 sustained minute following the tourniquet tape application. If no flow is observed for 1 sustained minute then the occlusion is considered successful. A still image is then saved for later evaluation by the blinded outcome assessor.
- Pneumatic Tourniquet: Automatic pneumatic tourniquet with a 10 cm (4 inch) wide cuff applied to the upper half of the participants thigh. Duplex and color flow ultrasound are used to assess distal blood flow at the popliteal artery for 1 sustained minute following the tourniquet tape application. If no flow is observed for 1 sustained minute then the occlusion is considered successful. A still image is then saved for later evaluation by the blinded outcome assessor.
- One Windlass Tourniquet: Duplex and color flow ultrasound are used to assess distal blood flow at the popliteal artery for 1 sustained minute following the application of a one windlass tourniquet to the middle upper thigh. If no flow is observed for 1 sustained minute then it is considered successful occlusion. A still image is then saved for later evaluation by the blinded outcome assessor.
- Two Windlass Tourniquets: Duplex and color flow ultrasound are used to assess distal blood flow at the popliteal artery for 1 sustained minute following the application of two windlass tourniquets to the middle upper thigh. If no flow is observed for 1 sustained minute then it is considered successful occlusion. A still image is then saved for later evaluation by the blinded outcome assessor.
Arm/Group | Tourniquet Tape 10 cm | Pneumatic Tourniquet | One Windlass Tourniquet | Two Windlass Tourniquets
Number analyzed (Participants) | 19 | 18 | 18 | 10
Participants
  Success: Absent flow verified by radiologist. | 19 | 18 | 8 | 8
  Failure: Flow verified by radiologist. | 0 | 0 | 10 | 2
Statistical Analysis 1: Comparison: Tourniquet Tape 10 cm vs One Windlass Tourniquet; Null hypothesis is that one windlass tourniquet is just as likely to occlude arterial flow as the 10 cm wide tourniquet tape. Participant count of 18 to accommodate for missing windlass tourniquet ultrasound data; Test type: Superiority or Other; p = 0.002, McNemar — Significance thresh hold: 0.05
Statistical Analysis 2: Comparison: One Windlass Tourniquet vs Two Windlass Tourniquets; Null hypothesis is that one windlass tourniquet is just as likely to occlude arterial flow as two windlass tourniquets. Participant count of 18 to accommodate for missing windlass tourniquet ultrasound data; Test type: Superiority or Other; p = 0.008, McNemar — Significance thresh hold: 0.05
Statistical Analysis 3: Comparison: Tourniquet Tape 10 cm vs Two Windlass Tourniquets; Null hypothesis is that the 10 cm wide tourniquet tape is just as likely to occlude arterial flow as using two windlass tourniquets. Participant count of 18 to accommodate for missing windlass tourniquet ultrasound data; Test type: Superiority or Other; p = 0.5, McNemar — Significance thresh hold: 0.05
Statistical Analysis 4: Comparison: Pneumatic Tourniquet vs Two Windlass Tourniquets; Null hypothesis is that using the pneumatic tourniquet is just as likely to occlude arterial flow as using two windlass tourniquets. Participant count of 17 to accommodate for missing ultrasound data; Test type: Superiority or Other; p = 0.5, McNemar — Significance thresh hold: 0.05

2. Primary Outcome: Investigator Limb Occlusion Assessment
Description: Duplex and color flow ultrasound are used to assess distal blood flow at the popliteal artery for 1 sustained minute following the application of each tourniquet intervention to the middle upper thigh. If no flow is observed for 1 sustained minute then it is considered a successful occlusion. This assessment was made by the investigator and ultrasonographer applying the intervention.
Time Frame: For 1 sustained minute after application of each tourniquet intervention.
Measure: Count of Participants; unit: Participants
Groups:
- Tourniquet Tape 10 cm: Tourniquet Tape 10 cm (4 inch) width. Duplex and color flow ultrasound are used to assess distal blood flow at the popliteal artery for 1 sustained minute following the tourniquet tape application. If no flow is observed for 1 sustained minute then the occlusion is considered successful.
- Pneumatic Tourniquet: Automatic pneumatic tourniquet with a 10 cm (4 inch) wide cuff applied to the upper half of the participants thigh. Duplex and color flow ultrasound are used to assess distal blood flow at the popliteal artery for 1 sustained minute following the tourniquet tape application. If no flow is observed for 1 sustained minute then the occlusion is considered successful.
- One Windlass Tourniquet: Duplex and color flow ultrasound are used to assess distal blood flow at the popliteal artery for 1 sustained minute following the application of one windlass tourniquet to the middle upper thigh. If no flow is observed by the investigators for 1 sustained minute then it is considered successful occlusion.
- Two Windlass Tourniquets: Duplex and color flow ultrasound are used to assess distal blood flow at the popliteal artery for 1 sustained minute following the application of the two windlass tourniquets to the middle upper thigh. If no flow is observed by the investigators for 1 sustained minute then it is considered successful occlusion.
- Tourniquet Tape 5 cm: Tourniquet Tape 5 cm (2 inch) width. Duplex and color flow ultrasound are used to assess distal blood flow at the popliteal artery for 1 sustained minute following the tourniquet tape application. If no flow is observed for 1 sustained minute then the occlusion is considered successful.
Arm/Group | Tourniquet Tape 10 cm | Pneumatic Tourniquet | One Windlass Tourniquet | Two Windlass Tourniquets | Tourniquet Tape 5 cm
Number analyzed (Participants) | 19 | 19 | 19 | 11 | 4
Participants
  Success: Absent flow observed by investigator. | 19 | 19 | 8 | 9 | 3
  Failure: Flow observed by investigator. | 0 | 0 | 11 | 2 | 1

ADVERSE EVENTS:
Time Frame: 1 day
Groups:
- Pneumatic Tourniquet: The Automatic Tourniquet System (ATS) 1500 by Zimmer (formerly Aspen Labs) was used with a 10 cm (4 inch) wide pneumatic cuff.
- Windlass Tourniquet: One or two windlass tourniquets applied as needed to achieve study objectives.
- Tourniquet Tape 5 cm: Tourniquet Tape 5 cm (2 inch) width. A highly elastic transparent occlusive material that can create circumferential pressure when stretched and wrapped around a limb.
- Tourniquet Tape 10 cm: Tourniquet Tape, 10 cm (4 inch) width. A highly elastic transparent occlusive material that can create circumferential pressure when stretched and wrapped around a limb.
Arm/Group | Pneumatic Tourniquet | Windlass Tourniquet | Tourniquet Tape 5 cm | Tourniquet Tape 10 cm
All-Cause Mortality (participants affected / at risk) | 0/19 | 0/19 | 0/4 | 0/19
Serious Adverse Events (participants affected / at risk) | 0/19 | 0/19 | 0/4 | 0/19
Other Adverse Events (participants affected / at risk) | 0/19 | 0/19 | 0/4 | 0/19

LIMITATIONS AND CAVEATS:
Tourniquet tape 5 cm ended early due to excessive narrowing, resulting in data loss.

The pressure mapping system proved subjective in use and software bugs resulted corrupt data files.

Small sample size, therefore only large individuals enrolled.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No